CLINICAL TRIAL: NCT04722107
Title: Safety Trial of rAAV2/8-hCYP4V2 Gene Replacement Therapy Drug Administered as a Single Subretinal Injection in Patients With Bietti's Crystalline Dystrophy (BCD)
Brief Title: Safety Study of rAAV2/8-hCYP4V2 in Patients With Bietti's Crystalline Dystrophy (BCD)
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZVS101e-01
Record Dates: First submitted 2021-01-11; First posted 2021-01-25 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2022-07

CONDITIONS: Bietti's Crystalline Dystrophy
MeSH Terms: conditions — Bietti Crystalline Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): All patients enrolled in the study will receive a single subretinal injection of ZVS101e in one eye
  Interventions: Drug: rAAV2/8-hCYP4V2

INTERVENTIONS:
Drug: rAAV2/8-hCYP4V2 — rAAV2/8-hCYP4V2 is developed by Chigenovo Co., Ltd., it contains recombinant adeno-associated virus serotype 8 (rAAV8) vectors which carry human CYP4V2 gene
  Other Names: ZVS101e; rAAV8-hCYP4V2

SUMMARY:
Primary Objectives: To evaluate the safety of rAAV2/8-hCYP4V2 gene replacement therapy drug administered as a single subretinal injection in patients with Bietti's Crystalline Dystrophy (BCD).

Secondary Objectives: To preliminarily explore the clinical effectiveness of rAAV2/8-hCYP4V2 gene replacement therapy drugs.

DETAILED DESCRIPTION:
This is a single-arm, open-label, and single-center study of ZVS101e in patients with BCD. A total of 12 participants will be enrolled. A retinal surgeon will administer the vector by subretinal injection. Safety, efficacy and vector shedding characteristics of ZVS101e are then measured over 2 years.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥ 18 years old at the time of informed consent ;
* 2) Patients with a clinical diagnosis of Bietti's crystalline dystrophy (BCD);
* 3) Genetic test confirmed to carry two pathogenic variants of CYP4V2;
* 4) Meet the following target eye selection criteria： Best corrected visual acuity between 2.3 LogMAR and 0.5 LogMAR (including 2.3 LogMAR and 0.5 LogMAR, equivalent to Snellen visual acuity of hand move to 20/63); No refractive media clouding affecting fundus examination, visual examination and retinal function examination; The eye with the poorer visual acuity of the two eyes of the subject is the target eye. Note: For all subjects, only one eye will be used as the "target eye". If both eyes meet the inclusion criteria and the visual acuity is comparable, the target eye will be determined medically by the investigator.
* 5) Agree to take effective contraceptive measures from the beginning of the study to 2 year after the administration;
* 6) Voluntarily participate in this clinical trial and have signed the informed consent form.

Exclusion Criteria:

* 1) Patients lack sufficient retinal photoreceptors, retinal photoreceptors less than 1 optic disc area or retinal thickness less than 100 μm in the macula；
* 2) Existing or pre-existing of choroidal neovascular (CNV) lesions that were secondary to BCD, or other eye conditions interfering（ (e.g., high refractive error, retinal vasculitis, etc.) ） that may prevent surgery or interfere with the interpretation of the study endpoint;
* 3) Prior use of medicines which may affect the experimental observation within the 6 months before screening (such as ranibizumab, bevacizumab, aflibercept, conbercept)；
* 4) Prior intraocular surgery in the target eye (e.g. PDT, pars plana vitrectomy, retinal laser therapy )
* 5) Currently taking or may require systemic medications that can cause ocular toxicity, such as psoralen, risedronate, or tamoxifen；
* 6) Allergic constitution (such as those who are allergic to two or more drugs and foods);
* 7) Abnormal physical examination, vital signs, laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function, immunological examination, female blood pregnancy), 12-lead ECG, X-ray chest radiograph findings with any clinically significant abnormality, and where participation in this study may increase the subject's risk or interfere with data interpretation as assessed by the investigator；
* 8) Having any past or present medical history that may affect the safety of the trial or the in vivo process of the drug, especially the medical history of cardiovascular, hepatic, renal, endocrine, gastrointestinal, pulmonary, neurological, hematological, oncologic, immunological or metabolic disorders and others that are thought clinically significant by the investigator；
* 9) Participation in any medicine or medical device clinical trials within 3 months prior to enrollment;;
* 10) Neutralizing antibodies to rAAV> 1:1000 by immunologic test;
* 11) For females in pregnancy or lactation period;
* 12)Carrying other ophthalmic pathogenic mutations
* 13) Any other conditions which leads the investigator to determine the participant is unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2024-01-25 (Estimated); Study Completion 2024-04-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 24 months
  Incidence of adverse events, vital signs, physical examination, ophthalmic An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event will not need to have a causal relationship with the treatment.
Incidence of serious adverse events | 24 months
  A serious adverse event (SAE) is any untoward medical occurrence at any dose that leading to the following:
  Results in death; Life-threatening, refers to an event in which the patient is at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe; Significant or permanent disability/incapacity, where disability refers to a serious disruption and damage of a person's ability to perform normal life functions; Requires inpatient hospitalization or prolongation of existing hospitalization; Congenital anomaly or birth defect; Other medically important events
Clinically important changes from baseline after ZVS101e treatment | 24 months
  Clinically important changes including abnormal physical examinations, vital signs, ECG, laboratory findings (chemistry, hematology, urinalysis) and ophthalmologic findings (BCVA, slit lamp examination, ophthalmoscopy, IOP, funds photography, FAF, OCT, OCTA).

SECONDARY OUTCOMES:
Mean change from baseline in BCVA after ZVS101e treatment | 24 months
  BCVA of both eyes will be assessed using the early treatment of diabetic retinopathy study (ETDRS) chart
Change from Baseline in visual field | 24 months
  Visual field will be assessed by Humphrey perimetry, changes in VFI, MD, PSD will be analyzed.
Change from Baseline in contrast sensitivity | 24 months
  Change from baseline in contrast sensitivity will be measured using the CSV-1000E instrument.
Change from Baseline in multi-luminance mobility test (MLMT) | 24 months
  MLMT was assessed at 1 or more of 7 levels of illumination, ranging from 400 lux (a brightly lit office) to 1 lux (a moonless summer night). The score range is between -1 (the worst) and 6 (the best).
Change from Baseline in OCTA | 24 months
  The OCTA examines the retinal and choroidal vessels. The retinal and choroidal vessel perfusion area, vessel volume, and vessel index will be analyzed.
Change from Baseline in microperimetry | 24 months
  Microperimetry will be measured using MP-3，changes in retinal light sensitivity will be analyzed.
Change from Baseline in mfERG | 24 months
  The measurement will be performed based on the standards of international society for clinical electrophysiology of vision (ISCEV).The change of retinal function in the macula will be analyzed.
Change from Baseline in retinal thickness | 24 months
  Retinal thickness will be assessed for both eyes using OCT.
Change from Baseline in NEI VFQ-25 total score | 24 months
  National eye institute 25-item visual function questionnaire (NEI VFQ-25) consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively.
Change from Baseline in fundus autofluorescence (FAF) | 24 months
  FAF is a noninvasive test to explore the health and metabolic status of retinal pigment epithelial cell/photoreceptor complex.

CONTACTS AND LOCATIONS:
Overall Officials: wenbin Wei, Doctor, Principal Investigator — Vice President of Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jia R, Meng X, Chen S, Zhang F, Du J, Liu X, Yang L. AAV-mediated gene-replacement therapy restores viability of BCD patient iPSC derived RPE cells and vision of Cyp4v3 knockout mice. Hum Mol Genet. 2023 Jan 1;32(1):122-138. doi: 10.1093/hmg/ddac181. PMID 35925866